CLINICAL TRIAL: NCT01818518
Title: Neonatal Outcome by Reason for Delivery - A Prospective, Observational Study
Brief Title: Neonatal Outcome by Reason for Delivery
Status: Completed | Type: Observational
Sponsor: Obstetrix Medical Group (Industry)
Responsible Party: Sponsor
Organization: Pediatrix (Other)
Other Study IDs: OBX0022
Record Dates: First submitted 2013-03-21; First posted 2013-03-26 (Estimated); Results first posted 2019-06-07 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Preterm Delivery
Keywords: Preterm delivery; Premature delivery; Premature birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Preterm Labor: Group who goes into labor prior to 32 weeks of gestation
- Prelabor rupture of membranes: Group who have prelabor rupture of membranes are those who break their bag of water prior to 32 weeks gestation in the absence of labor.
- Premature birth before 32 weeks gestation: Premature birth before 32 weeks gestation not including PTL or PROM

SUMMARY:
To determine the rate of Composite Neonatal Morbidity for very preterm babies delivered secondary to preterm labor (PTL) vs. prelabor rupture of membranes (PROM). Composite neonatal morbidity is defined as ≥ 1 of the following: Respiratory Distress Syndrome (RDS) (oxygen requirement, clinical diagnosis, and consistent chest radiograph), bronchopulmonary dysplasia (BPD) (requirement for oxygen support at 28 days of life), severe intraventricular hemorrhage (IVH) (grades III or IV), periventricular leukomalacia (PVL), blood culture-proven sepsis, necrotizing enterocolitis (NEC), or perinatal death (stillbirth or death before neonatal hospital discharge.

DETAILED DESCRIPTION:
This is a prospective, observational study that will use information from the medical records of mothers and their newborns. This study seeks to determine the rate of Composite Neonatal Morbidity for very preterm babies delivered secondary to preterm labor (PTL) vs. prelabor rupture of membranes (PROM). Composite neonatal morbidity is defined as ≥ 1 of the following: Respiratory Distress Syndrome (RDS) (oxygen requirement, clinical diagnosis, and consistent chest radiograph), bronchopulmonary dysplasia (BPD) (requirement for oxygen support at 28 days of life), severe intraventricular hemorrhage (IVH) (grades III or IV), periventricular leukomalacia (PVL), blood culture-proven sepsis, necrotizing enterocolitis (NEC), or perinatal death (stillbirth or death before neonatal hospital discharge.

Secondary Objectives: 1) Difference in mortality between the PTL and PROM groups, composite morbidity differences for other reasons for premature delivery, and individual morbidities including IVH, PVL, RDS, sepsis, seizures, BPD and NEC

Study Population: All babies from singleton pregnancies delivering in each of the involved hospitals who deliver at less than 32 weeks of gestation who are stillborn, who die in the delivery room and who are cared for in the Neonatal Intensive Care Unit (NICU) will be included.

Planned Sample Size: We plan a two year study and estimate based on historical data for the institutions to be included in the study, which should yield approximately 6000 babies less than (<) 32w0d gestation. For a 10% difference in composite morbidity (assuming 90% power and two-sided alpha=0.05) assuming a rate of 60% at least 661 patients are needed in each of the 3 groups (PTL, PROM, and other).

ELIGIBILITY:
Inclusion Criteria:

* Delivery at participating hospitals at less than 32weeks of gestation based on best obstetrical dating
* Singleton pregnancy
* Delivery where the baby is:

  1. Stillborn OR
  2. Born alive and:
* expires before it leaves the delivery room OR
* is cared for in the Neonatal Intensive Care Unit or an Intermediate Care Nursery

Exclusion Criteria:

* Patient less than 18 years of age
* Pregnancies that had previously been multiple gestations but where one or more fetuses had died after 12weeks of gestation
* Deliveries where the baby is born alive, does not expire in the delivery room but the baby does not get admitted to the NICU.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All babies from singleton pregnancies delivering in each of the involved hospitals who delivered at less than 32 weeks of gestation and who are stillborn, who die in the delivery room and who are cared for in the Neonatal Intensive Care Unit (NICU) will be included.
Sampling Method: Non-Probability Sample
Enrollment: 995 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2016-05-03 (Actual); Study Completion 2016-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Garite, MD, Principal Investigator — Obstetrix Medical Group
Locations (10):
- United States (10):
  - Banner Desert Medical Center, Mesa, Arizona
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - Scottsdale Healthcare-Shea Medical Center, Scottsdale, Arizona
  - Saddleback Memorial Medical Center, Laguna Hills, California
  - Good Samaritan Hospital, San Jose, California
  - Presbyterian/St Luke's Hospital, Denver, Colorado
  - Saint Luke's Hospital, Kansas City, Kansas City, Missouri
  - Mercy Hospital of St. Louis, St Louis, Missouri
  - Harris Methodist Hospital - Fort Worth, Fort Worth, Texas
  - Swedish Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided
undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Prelabor Rupture of Membranes Diagnosis on Admission: Group who have prelabor rupture of membranes (PROM) are those who break their bag of water prior to 32 weeks gestation in the absence of labor. Diagnosis made on admission
- Preterm Labor Diagnosis on Admission: Group who goes into labor prior to 32 weeks of gestation. Diagnosis was made on admission
- Pre-eclampsia Diagnosis on Admission: The diagnosis of Preeclampsia at time of admission
- Intrauterine Growth Restriction (IUGR) Diagnosis on Admission: The diagnosis of IUGR at time of admission
- Vaginal Bleeding Diagnosis on Admission: The diagnosis of vaginal bleeding made at time of admission
- Short Cervix Diagnosis on Admission: The diagnosis of Short cervical length at time of admission
Period: Overall Study
Arm/Group | Prelabor Rupture of Membranes Diagnosis on Admission | Preterm Labor Diagnosis on Admission | Pre-eclampsia Diagnosis on Admission | Intrauterine Growth Restriction (IUGR) Diagnosis on Admission | Vaginal Bleeding Diagnosis on Admission | Short Cervix Diagnosis on Admission
Started | 310 | 263 | 288 | 59 | 38 | 37
Completed | 310 | 263 | 288 | 59 | 38 | 37
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- IUGR Diagnosis on Admission: The diagnosis of IUGR at time of admission
- Total: Total of all reporting groups
Arm/Group | Prelabor Rupture of Membranes Diagnosis on Admission | Preterm Labor Diagnosis on Admission | Pre-eclampsia Diagnosis on Admission | IUGR Diagnosis on Admission | Vaginal Bleeding Diagnosis on Admission | Short Cervix Diagnosis on Admission | Total
Number analyzed (Participants) | 310 | 263 | 288 | 59 | 38 | 37 | 995
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.7 (6.0) | 28.1 (6.0) | 29.9 (6.5) | 28.6 (5.6) | 28.9 (6.2) | 29.4 (5.6) | 29.1 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 310 | 263 | 288 | 59 | 38 | 37 | 995
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Participants were able to indicate more than one Race/Ethnicity in their response. Population: Not all ethnicity data was available for all participants enrolled in the study and participants were able to select more than one Race/Ethnicity when applicable.
  Participants
    White: number analyzed (Participants) | 299 | 257 | 284 | 59 | 36 | 36 | 971
    White | 163 | 139 | 142 | 33 | 21 | 19 | 517
    Hispanic: number analyzed (Participants) | 299 | 257 | 284 | 59 | 36 | 36 | 971
    Hispanic | 67 | 51 | 61 | 9 | 4 | 5 | 197
    Black: number analyzed (Participants) | 299 | 257 | 284 | 59 | 36 | 36 | 971
    Black | 32 | 25 | 35 | 6 | 7 | 8 | 113
    Asian: number analyzed (Participants) | 299 | 257 | 284 | 59 | 36 | 36 | 971
    Asian | 11 | 18 | 13 | 3 | 3 | 2 | 50
    Other: number analyzed (Participants) | 299 | 257 | 284 | 59 | 36 | 36 | 971
    Other | 37 | 30 | 37 | 8 | 3 | 3 | 118
Region of Enrollment [Number; unit: participants]
  United States | 310 | 263 | 288 | 59 | 38 | 37 | 995
Nulliparity [Count of Participants; unit: Participants] — Population: number analyzed if different from total number because these characteristic were not captured on all patients. Some baseline data was unknown.
  Participants
    number analyzed (Participants) | 292 | 255 | 282 | 59 | 33 | 35 | 956
    (all) | 100 | 108 | 133 | 22 | 7 | 17 | 387
Prenatal Care [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: number analyzed if different from total number because these characteristic were not captured on all patients. Some baseline data was unknown
  Participants
    number analyzed (Participants) | 298 | 255 | 284 | 59 | 36 | 36 | 968
    (all) | 290 | 247 | 273 | 57 | 34 | 33 | 934
Gestational Age at admission , wks [Mean (Standard Deviation); unit: weeks] | 27.1 (2.7) | 27.7 (2.6) | 28.3 (2.2) | 28.2 (2.3) | 26.7 (2.9) | 24.4 (2.3) | 27.0 (2.5)
Gestational Age at delivery, wks [Mean (Standard Deviation); unit: weeks] | 28.5 (2.5) | 28.1 (2.5) | 28.9 (2.1) | 29.1 (2.2) | 27.4 (2.6) | 26.3 (2.6) | 28.1 (2.4)
Interval from admission to delivery, wks. [Mean (Standard Deviation); unit: weeks] | 1.4 (1.6) | 0.4 (0.7) | 0.6 (0.7) | 0.9 (1.1) | 0.7 (1.0) | 1.8 (2.0) | 1.0 (1.2)
Cesarean delivery [Count of Participants; unit: Participants] | 178 | 107 | 268 | 58 | 27 | 22 | 660
Received full course of antenatal corticosteroids [Count of Participants; unit: Participants] — A full course was determined by evaluation of the medical record to verify that two doses of antenatal corticosteroid prior to rupture of membranes and each dose was administered 24 hours apart.
  Participants | 138 | 114 | 195 | 32 | 14 | 19 | 512
Male newborn [Count of Participants; unit: Participants] | 178 | 149 | 145 | 33 | 22 | 24 | 551
Primary reason for delivery = spontaneous labor [Count of Participants; unit: Participants] | 171 | 228 | 0 | 2 | 11 | 21 | 433
Primary reason for delivery = preeclampsia [Count of Participants; unit: Participants] | 0 | 0 | 219 | 3 | 0 | 0 | 222
Primary reason for delivery = fetal heart rate nonreassuring [Count of Participants; unit: Participants] | 54 | 15 | 49 | 42 | 7 | 6 | 173
Primary reason for delivery = chorioamnionitis [Count of Participants; unit: Participants] | 54 | 12 | 0 | 0 | 0 | 5 | 71
Primary reason for delivery = Bleeding [Count of Participants; unit: Participants] | 18 | 6 | 8 | 0 | 20 | 1 | 53
Primary reason for delivery = Other [Count of Participants; unit: Participants] | 13 | 2 | 12 | 12 | 0 | 4 | 43

OUTCOME MEASURES:

1. Primary Outcome: Composite Perinatal Morbidity
Description: The primary outcome is Composite Perinatal Morbidity. Composite morbidity refers to the newborns born to the female participants enrolled in the study. Composite Morbidity is defined as ≥ 1 of the following: respiratory distress syndrome (RDS) (oxygen requirement, clinical diagnosis, and consistent chest radiograph), bronchopulmonary dysplasia (BPD) (requirement for oxygen support at 28 days of life), severe intraventricular hemorrhage (IVH) (grades III or IV), periventricular leukomalacia (PVL), blood culture-proven sepsis present within 72 hours of birth, necrotising enterocolitis (NEC), or perinatal death (stillbirth or neonatal death prior to hospital discharge).
Time Frame: Infants from birth until discharge or until infant reaches 28 days of life.
Population: Composite morbidity is defined as ≥ 1 of the following: RDS, BPD, severe IVH (grades III or IV), PVL, blood culture-proven sepsis present within 72 hours of birth, NEC, or perinatal death. Perinatal Morbidity assessed pertains to the newborns born to the enrolled female patients.
Measure: Number; unit: participants
Arm/Group | Prelabor Rupture of Membranes Diagnosis on Admission | Preterm Labor Diagnosis on Admission | Pre-eclampsia Diagnosis on Admission | IUGR Diagnosis on Admission | Vaginal Bleeding Diagnosis on Admission | Short Cervix Diagnosis on Admission
Number analyzed (Participants) | 310 | 263 | 288 | 59 | 38 | 37
participants
  Composite Morbidity | 277 | 203 | 221 | 45 | 28 | 33
  Serious Morbidity | 82 | 68 | 62 | 20 | 17 | 20
  Perinatal (infant) Death | 32 | 20 | 17 | 6 | 5 | 5
  Respiratory distress syndrome (RDS) | 206 | 190 | 211 | 43 | 23 | 27
  On Ventilatory at 28 days of age | 24 | 28 | 29 | 14 | 11 | 10
  Intraventicular Hemorrhage Grade 3 or 4 | 13 | 19 | 8 | 1 | 5 | 8
  Necrotizing Enterocolitis | 9 | 15 | 14 | 3 | 5 | 2
  Periventricular Leukomalacia (PVL) | 2 | 1 | 1 | 1 | 1 | 0
  Sepsis | 11 | 5 | 6 | 2 | 1 | 1
  Cord arterial pH < 7.1 | 8 | 7 | 14 | 2 | 5 | 0
  Cord venous pH <7.1 | 5 | 5 | 9 | 2 | 3 | 0
  Arterial base excess < -12 | 5 | 3 | 6 | 1 | 2 | 0
  Venous Base Excess < -12 | 2 | 4 | 5 | 1 | 2 | 0
  Five-minute Apgar score < 5 | 24 | 15 | 15 | 2 | 2 | 6

ADVERSE EVENTS:
Time Frame: No adverse events were assessed from the beginning through the duration of the study. This is an observational study and therefore adverse events were not assessed.
Description: All-Cause Mortality, Serious, and Other Adverse Events were not monitored/assessed in this observational study.
Groups:
- IUGR Diagnosis on Admission: Group who have the diagnosis of intrauterine growth restriction on admission to the hospital.
- Pre-Eclampsia Diagnosis on Admission: Group who have the diagnosis of pre-eclampsia noted on admission to the hospital
- Vaginal Bleeding Diagnosis on Admission: Group who have the presence of vaginal bleeding noted at the time of admission to the hospital
- Short Cervix Diagnosis on Admission: Group who have the diagnosis of a short cervical length at the time of admission to the hospital
Arm/Group | Preterm Labor | Prelabor Rupture of Membranes | IUGR Diagnosis on Admission | Pre-Eclampsia Diagnosis on Admission | Vaginal Bleeding Diagnosis on Admission | Short Cervix Diagnosis on Admission
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes